CLINICAL TRIAL: NCT03139500
Title: A Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-61803534 and an Open-Label Study to Evaluate the Effect of JNJ-61803534 on the Pharmacokinetics of Midazolam in Healthy Participants
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-61803534 and to Evaluate the Effect of JNJ-61803534 on the Pharmacokinetics of Midazolam in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to nonclinical findings
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108320; 2016-004085-26 (EudraCT Number); 61803534NAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will receive single oral doses of JNJ-61803534 or placebo in the fasted or fed state.
  Interventions: Drug: JNJ-61803534; Drug: Placebo
- Part 2: Multiple Ascending Dose (MAD) (Experimental): Participants will receive JNJ-61803534 or placebo over a 14-day period.
  Interventions: Drug: JNJ-61803534; Drug: Placebo
- Part 3: Drug-drug Interaction (DDI) (Experimental): Participants will receive single oral doses of midazolam on Day 1 and Day 16 and will receive JNJ-61803534 daily from Day 3 through Day 16 for 14 days at a dose based on the data from the SAD and MAD part.
  Interventions: Drug: JNJ-61803534; Drug: Midazolam

INTERVENTIONS:
Drug: JNJ-61803534 — Participants will receive JNJ-61803534 tablets orally.
Drug: Placebo — Participants will receive matching placebo.
  Arms: Part 1: Single Ascending Dose (SAD); Part 2: Multiple Ascending Dose (MAD)
Drug: Midazolam — Participants will receive single oral dose of midazolam.
  Arms: Part 3: Drug-drug Interaction (DDI)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and pharmacokinetics of JNJ61803534 in healthy participants after administration of single ascending oral doses of JNJ-61803534 (Part 1) and multiple ascending oral doses of JNJ-61803534, administered for 14 consecutive days (Part 2) as well as the potential of JNJ-61803534 to interact with other drugs (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) (BMI = weight/height^2), and a body weight of not less than 50 kilogram (kg)
* Participant must be healthy on the basis of their medical history, a physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed during screening
* Participant must be healthy on the basis of clinical laboratory tests performed during screening and at Day -1
* A woman must have a negative urine pregnancy test at screening and a negative highly sensitive serum pregnancy test on Day -1

Exclusion Criteria:

* Participant has a history of liver or renal insufficiency or significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, dermatologic, rheumatologic, psychiatric, or metabolic disturbances
* Participant has a history of malignancy before screening. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk of recurrence
* Participant has an active acute or chronic infection (including chronic recurrent or invasive candidiasis) or diagnosed latent infection
* Participant has received an investigational treatment (including investigational vaccines) within 2 months or 5 half-lives (whichever is longer) or used an invasive investigational medical device within 3 months before the planned first dose of study treatment or is currently enrolled in an investigational study
* Participant had major surgery, (example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study or within 4 weeks after the last dose of study treatment administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) as a Measure of Safety: Part 1 | Approximately up to 12 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Percentage of Participants With AEs as a Measure of Safety: Part 2 | Approximately up to 14 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-61803534 (Parts 1, 2 and 3) | Pre-dose, up to Day 50 (Part 1), up to Day 60 (Part 2), and up to Day 63 (Part 3)
  Plasma concentration assessment will be done to characterize the pharmacokinetics (PK) of of JNJ-61803534.
Plasma Concentration of Midazolam (Part 3) | Pre-dose and up to Day 18
  Plasma concentration assessment will be done to characterize the effect of JNJ-61803534 on the PK of midazolam.
Inhibition of Stimulated IL-17A Production in Diluted Whole Blood (Parts 1 and 2) | Pre-dose, up to Day 22 (Part 1 - SAD) and up to Day 43 (Part 2 - MAD)
  The amount of IL-17A secreted during the ex-vivo stimulation will be measured during the dosing period.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium